CLINICAL TRIAL: NCT03460470
Title: Sildenafil in US Heart Failure Patients (SilHF-US)
Acronym: SilHF-US
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Konstadina Darsaklis, MD, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHC-2016-0152
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil 40mgx3 daily (Active Comparator): Sildenafil 40mgx3 daily for 6 months
  Interventions: Drug: Sildenafil
- Placebo tablet x3 daily (Placebo Comparator): Placebo for Sildenafil 40mgx3 daily for 6 months
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Sildenafil — PDE5 Inhibitor
  Arms: Sildenafil 40mgx3 daily
Drug: Placebo oral capsule — Placebo for Sildenafil
  Arms: Placebo tablet x3 daily

SUMMARY:
This protocol describes a 2-arm randomized controlled pilot study assessing the tolerance, safety and efficacy of sildenafil compared to control. The hypothesis is that sildenafil will be well tolerated and efficacious in patients with chronic heart failure (NYHA class II and III) with evidence of systolic dysfunction (EF ≤40 %) and secondary pulmonary hypertension (SPAP >40mmHg).

Patients that satisfy the inclusion criteria will be randomized to sildenafil (40mg x 3) or placebo therapy for 6 months in a 2:1 blinded fashion. The placebo group will be compared to the active therapy group and analyzed for differences in the main study end-points Patient Global Assessment and 6-Minute Walk Test.

The study will also assess safety, tolerability, symptoms and quality of life.

DETAILED DESCRIPTION:
It is estimated that 2-3 % of the adult population suffers from heart failure (HF) and the prevalence is increasing. The European Society of Cardiology (ESC) represents countries with a population > 1,1 billion, and it is estimated that approximately 30 million patients have HF in these 53 countries. Heart failure is particularly prevalent in the elderly population and represents a major burden for both patients and the health services. In United states (US) more than 5 million people, or almost 2% of population have HF (Go at al, 2013) Medicare data indicate that 12% to 27% of patients hospitalized for heart failure are readmitted within 30 days after their discharge, and all-cause mortality reaches 12% in the same period. (Jencks at al, 2009).

Despite optimal non-pharmacological, pharmacological and device therapy, the morbidity among HF patients is high with symptoms such as dyspnoea and fatigue that reduce quality of life. Following diagnosis approximately 50% are dead after 4 years. Forty percent of patients admitted to hospital with HF are either dead or hospitalized within one year.

During the last decade, PDE5-inhibitors have been evaluated as a potential treatment for heart failure (see scientific rationale and reference). However, these investigations have been small and there is still limited data. Trials assessing the acute effects of PDE5-inhibition in patients with symptomatic HF due to systolic dysfunction have been performed primarily with sildenafil. Due to the short half-life of sildenafil the drug is administered 3 times daily when studying its chronic effects.

Previous studies have evaluated the 50 mg dose acutely and 50 mg 3 times daily during short-term chronic studies. Importantly, there is considerable off-label use of sildenafil in symptomatic heart failure patients in most European countries.

Revatio is currently licensed for pulmonary hypertension group 1. The dosing scheme is 20mg x 3. However, we suggest targeting a higher dose to achieve optimal clinical benefit in patients with heart failure and moderate congestion. As mentioned above most of the clinical literature in patients with symptomatic heart failure has been done using the 50mg x 3 regimen. However, it is believed that in the proposed study using 40mg x 3 should be equally efficacious. There is already considerable experience using this dosage scheme in heart failure patients locally.

The hemodynamic profile of PDE-5 inhibitors is favorable with reduction in filling pressures, both systemic and pulmonary, vascular resistance accompanied by improvement in symptoms and sub maximal and peak exercise performance. This pilot study will evaluate the use of the PDE5-inhibitor sildenafil in patients with heart failure, systolic dysfunction and documented secondary pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. 18 - 80 years of age.
3. Outpatients with chronic HF. NYHA class II-III on optimal treatment in sinus rhythm or atrial fibrillation
4. LVEF ≤ 40% measured during the past 12 months
5. SPAP ≥ 40mmHg using echocardiography
6. 6MWTD < 475 meters
7. NT-pro BNP ≥ 400 pg/ml or BNP ≥100 pg/ml, measured during the past 12 months
8. Receiving optimal therapy, including diuretic, ACE-inhibitor, ARB, beta-blocker and aldosterone antagonist. Doses of all medication should be unchanged during the last 30 days before inclusion.
9. ICDs and CRTs (CRT-P, CRT-D) are permitted. Implantation should have been performed at > 3 months before inclusion to the trial.

Exclusion Criteria: -

1. Acute Coronary Syndrome, including myocardial infarction, or coronary angiography, with or without intervention, within the last 3 months
2. Stroke within the last 3 months
3. Planned coronary angiography or planned device-implantation
4. Moderate to severe obstructive valve disease
5. Documented episodes of sustained ventricular tachycardia
6. Prior (past 30 days before the baseline visit) or ongoing use of oral nitrate therapy.
7. Concomitant disease which interfere with assessment of dyspnea , severe COPD, asthma, restrictive lung disease, severe obesity
8. Anemia (hemoglobin < 10g/dL)
9. Uncontrolled hypertension ( SBP >160 mmHg and / or DBP > 90 mmHg)
10. Symptomatic or orthostatic hypotension or systolic blood pressure < 90 mmHg
11. Clinically important renal dysfunction (GFR < 40m ml/min)
12. Women with child-bearing potential
13. Prior (past 30 days before the baseline visit) or ongoing use of i) alpha-1 antagonist: doxazosin ii) CYP3A4 inhibitors: erytromycin, ritonavir, sakinovir, itrakonazole, ketokonazole iii) CYP3A4-inducers: rifampicin iv) Any calcium channel blockers
14. V) Pulmonary vasodilators at the treatment dose level for Pulmonary hypertensionRetinitis pigmentosa, previous diagnosis of NAION (non-arteritic ischemic opticus-neuropathy), unexplained visual disturbance.
15. Sickle cell anemia, multiple myeloma, leukemia or penile anatomic deformities (angulation, cavernosal fibrosis, Peyronie's disease) that increases the risk of priapism.
16. Hepatic failure.
17. Drug and alcohol abuse which precludes compliance with the protocol.
18. Inability to understand or sign the written informed consent form of the study,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Six minute walk test | Baseline, 8 weeks and 24 weeks
  Analysis of change from the baseline
Patient Global Assessment (PGA) | Baseline; 8 weeks and 24 weeks
  Analysis of change form the baseline

SECONDARY OUTCOMES:
1.Quality of Life (QoL) evaluation by EuroQol5D | Baseline, 8 weeks and 24 weeks
  Analysis of change from baseline
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, 8 weeks and 24 weeks
  Analysis of change from baseline
New York Heart Association (NYHA) function class | Baseline, 8 weeks and 24 weeks
  Analysis of change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Konstadina Darsaklis, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital 80 Seymour street, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
The SilHF trial is an international, multi-centre effort with five participating European centres.The Steering Committee of the SilHF trial, has elected to pool the individual patient data from the five European centers with a large single center in Hartford Connecticut, USA, PI: Konstadina Darsaklis. The US site will follow an identical protocol to the European sites and enter data on the electronic case report form to the data management centre in Trondheim, Norway. We intend to perform the meta-analysis independent of the results of the separate studies. All sites have obtained the required regulatory approvals.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The only US site at Hartford Hospital will complete enrollment by the end of year 2018. Data will be available and study database will be updated within 5 days of any obtained f-u visit.
Access Criteria: De-identified coded data will be entered into a secure login study database.

REFERENCES:
- [Result] Guazzi M, Dickstein K, Vicenzi M, Arena R. Six-minute walk test and cardiopulmonary exercise testing in patients with chronic heart failure: a comparative analysis on clinical and prognostic insights. Circ Heart Fail. 2009 Nov;2(6):549-55. doi: 10.1161/CIRCHEARTFAILURE.109.881326. Epub 2009 Sep 28. PMID 19919979
- [Result] Cooper TJ, Guazzi M, Al-Mohammad A, Amir O, Bengal T, Cleland JG, Dickstein K. Sildenafil in Heart failure (SilHF). An investigator-initiated multinational randomized controlled clinical trial: rationale and design. Eur J Heart Fail. 2013 Jan;15(1):119-22. doi: 10.1093/eurjhf/hfs152. Epub 2012 Oct 24. PMID 23097067